CLINICAL TRIAL: NCT04808258
Title: Value of Transthoracic Echocardiography and Long-term Holter Monitoring Following Embolic Stroke of Undetermined Source Detected by Magnetic Resonance Imaging: A Prospective Clinical Study
Brief Title: Embolic Stroke of Undetermined Source, Continuous Electrocardiography and Transthoracic ECHOcardiography in Hospitalized Patients With Ischemic Stroke
Acronym: ESECHO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Morten Lamberts, Associate Professor and Research Director, Herlev and Gentofte Hospital
Other Study IDs: H-20037212
Record Dates: First submitted 2021-02-21; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: transthoracic echocardiography; stroke; strain; embolism; secondary prevention
MeSH Terms: conditions — Stroke; Sprains and Strains; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C3+ Holter Monitor — Long-Term ECG monitoring (up to 7 days)

SUMMARY:
Transthoracic echocardiography (TTE) is recommended in patients with ischemic stroke when cardiac etiology is suspected to help plan secondary stroke management. However, discrepancy for specific clinical recommendation exists between cardiologists and neurologists, and data evaluating usefulness of TTE in unselected patients with cryptogenic strokes (CS) and embolic strokes of undetermined source (ESUS) are lacking. The investigators sought to evaluate the value of routinely performed echocardiography in consecutive CS/ESUS patients. The investigators will perform TTE as recommended by guidelines including agitated saline contrast and speckle-tracking to investigate potential implications for secondary stroke management. In addition, the researchers aim to evaluate the effectiveness of long-term continuous electrocardiogram (cECG) monitorering with newer Holter monitors to detect cardiac arrhythmia in patients with CS/ESUS.

In this prospective study, the investigators aim to evaluate 500 consecutive patients, regardless of age, in sinus rhythm with acute IS and potential cardioembolic stroke (CES) or cryptogenic stroke (CS/ESUS) according to Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria. Strokes are determined by magnetic resonance imaging. The researchers will perform TTE as recommended by guidelines including agitated saline contrast and speckle-tracking to investigate potential implications for secondary stroke management.

The investigators aim to explore underlying heart conditions and comorbidities among CES and ESUS patients. Data will include left atrium morphology, atrial septal aneurysm, valvular disease, mural thrombus and patent foramen ovale (PFO). Focus will be analysis of data on older patients, as some studies indicate that in ESUS patients >60 years of age, there is a higher prevalence of PFO in patients with low atherosclerosis and cardioembolic risk.

This project can potentially guide cardiologists and neurologists, on common grounds, for stroke management of potential cardioembolic origin. Implications of referring all-comers with stroke of potential cardioembolic origin to echocardiography will be illustrated.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with verified acute ischemic stroke determined by magnetic resonance imaging (MRI) and/or computed tomography (CT) of cerebrum.
* Patients, regardless of age, in sinus rhythm with acute IS and potential cardioembolic stroke or cryptogenic stroke (CS/ESUS) according to Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria.

Exclusion Criteria:

* Persons not able to cooperate.
* Persons unable to understand and sign "informed concent."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized patients with acute ischemic stroke from department of neurology (stroke unit) in University of Copenhagen Herlev Hospital.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-01-27 (Estimated); Study Completion 2022-03-27 (Estimated)

PRIMARY OUTCOMES:
Number (percentage) of patients with underlying heart conditions | 1 year
  Use of echocardiographic metrics (especially left atrial metrics) to guide secondary stroke management of patients suffering from embolic stroke of undetermined source (ESUS)..
Agreement in electrocardiogram findings between device A (new Holter monitor) and device B (traditional Holter monitor) | 1 year
  Use of long-term continuous electrocardiogram (cECG) monitoring with newer Holter monitors to detect cardiac arrhythmia and guide secondary stroke management of patients suffering from embolic stroke of undetermined source (ESUS)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Cardiology, Herlev & Gentofte Hospital, Copenhagen, Herlev
  - Department of Neurology, Herlev & Gentofte Hospital, Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: Undecided